CLINICAL TRIAL: NCT02465736
Title: A Phase III Clinical Trial of Docetaxel Plus Cisplatin Versus Vinorelbine Plus Cisplatin in Neoadjuvant Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma (NEOCRTEC308)
Brief Title: Study of Docetaxel or Vinorelbine Plus Cisplatin in Neoadjuvant Chemoradiotherapy for Esophageal Cancer (NEOCRTEC308)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOCRTEC-2.0
Record Dates: First submitted 2015-05-30; First posted 2015-06-08 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Cancer; Oesophageal Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Docetaxel; Cisplatin; Radiation; Surgical Procedures, Operative; Esophagectomy; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (DP-RT) (Experimental): • Arm A consists of the concurrent chemoradiotherapy prior to surgery. The patient will receive 4 weeks of radiation therapy and 4 weekly cycles of chemotherapy. The radiation will generally commence on the 1st day of treatment and will run for 4 weeks. Chemotherapy is given by intravenous infusion on days 1, 8, 15, and 22.
  Interventions:
  * Radiation: (44 Gy/20 fractions)
  * Drug: Docetaxel
  * Drug: Cisplatin
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: Radiation; Procedure: Surgery
- B (NP-RT) (Experimental): • Arm B consists of the concurrent chemoradiotherapy followed by surgery. The patient will receive 4 weeks of radiation therapy and 2 cycles of chemotherapy. The radiation will generally commence on the 1st day of treatment and will run for 4 weeks. Each cycle of chemotherapy lasts 21 days/3 weeks. The drugs include Vinorelbine and Cisplatin.
  Interventions:
  * Radiation: (44 Gy/20 fractions)
  * Drug: Vinorelbine
  * Drug: Cisplatin
  Interventions: Radiation: Radiation; Procedure: Surgery; Drug: Vinorelbine; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — 25mg/ m2 Docetaxel dose administered on days 1, 8, 15, and 22.
  Other Names: Docetaxel in Arm A
  Arms: A (DP-RT)
Drug: Cisplatin — 25mg/ m2 on days 1, 8, 15 and 22.
  Other Names: Cisplatin in Arm A
  Arms: A (DP-RT)
Radiation: Radiation — Patient will receive 4 weeks of radiation therapy (44 Gy/20 fractions).
  Other Names: IMRT
Procedure: Surgery — McKeown esophagectomy, Ivor Lewis esophagectomy or minimally invasive esophagectomy will be performed 4-8 weeks after chemoradiotherapy. Two-field lymphadenectomy with total mediastinal lymph node dissection is performed during surgery.
  Other Names: Esophagectomy
Drug: Vinorelbine — 25mg/ m2 on days 1, 8 of each cycle (i.e. every 21 days).
  Other Names: Vinorelbine in Arm B
  Arms: B (NP-RT)
Drug: Cisplatin — 75mg/ m2 on day 1 of each cycle only (i.e. every 21 days).
  Other Names: Cisplatin in Arm B
  Arms: B (NP-RT)

SUMMARY:
The primary objective is to compare docetaxel plus cisplatin (DP) versus vinorelbine plus cisplatin (NP) in neoadjuvant chemoradiotherapy, in terms of the overall survival and toxicity in patients with Stage IIB or III squamous cell esophageal carcinoma.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the eighth most common cancers in the world, with more than 456,000 new cases and 400,000 deaths occurred annually worldwide. Every year in China, no matter new cases or deaths account for more than half of the world. Besides, over 90% of Chinese patients have esophageal squamous cell carcinoma (ESCC).

Preoperative chemoradiotherapy (CRT) followed by surgery can hopefully improve the survival of ESCC. The CROSS trial has demonstrated that preoperative chemoradiotherapy can significantly increase the overall survival of patients with EC compared with surgery alone. The therapeutic effects were also found in 84 ESCC cases enrolled in this trial. Previously, the investigators performed a phase III, randomized clinical trial (NCT01216527) to compare the overall survival of stage IIB-III ESCC patients treated with or without neoadjuvant CRT, in which vinorelbine plus cisplatin was used as chemotherapy regime. The enrollment was completed in 2014. The outcomes will hopefully prove the survival benefit of neoadjuvant CRT to ESCC.

However, the investigators also observed that some patients suffer from the toxic response of neoadjuvant therapy, such as myelosuppression (45.2%), pulmonary toxicity (42.9%), and esophagitis (59.5%). The toxicity caused by CRT will decrease the patient compliance; moreover increase the perioperative complications and deaths, which may totally offset the survival benefit. Therefore, it is important to improve chemoradiotherapy effect and reduce toxicity, so as to achieve better survival in ESCC patients.

Docetaxel draws increasing attentions with its high effective rate and low toxicity. Several Phase II clinical trials and retrospective studies suggested that docetaxel showed better survival benefits in both monotherapy and combined-therapy in EC patients. Therefore, the investigators intended to conduct a phase III, randomized clinical trial to further explore whether docetaxel plus cisplatin would be an effective therapy with lower toxicity.

The investigators are to carry out a phased III clinical trial to compare the effect and toxicity of docetaxel plus cisplatin with vinorelbine plus cisplatin in neoadjuvant chemoradiotherapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage T1-4aN1-3M0 or T4aN0M0, according to 7th edition of Union for International Cancer Control (UICC) staging system.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival
4. Age ranges from 18 to 70 years
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. WHO performance status (PS) of 0-1
7. Signed informed consent document on file

Exclusion Criteria:

1. Patients have received any prior anticancer therapy
2. Patients with advanced inoperable or metastatic esophageal carcinoma
3. Patients with concomitant hemorrhagic disease
4. Patients with other uncontrollable status that cannot tolerate surgery
5. Pregnant or breast feeding
6. Patients cannot signed the informed consent document because of psychological quality, family and social factors
7. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more
8. Have a prior malignancy other than esophageal carcinoma, carcinoma in situ of the cervix, nonmelanoma skin cancer or cured early stage of prostate cancer
9. Have a history of diabetes over 10 years and with poorly controlled blood sugar level
10. patients with serious cardiac, respiratory, hepatic, renal, hematologic, immunological disease or cachexy, who cannot tolerate chemoradiotherapy or surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At end of trial- up to 3 years in follow up
  Overall survival will be calculated from the date of randomisation and an event registered on the date of death from any cause. Patients lost to follow up, or those with no death recorded on the day the database is frozen, will be censored on the date of last follow up.
Toxicities of neo-adjuvant chemoradiotherapy | Within the first 56 days after the start of chemoradiotherapy
  All symptoms of toxicity will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) Version. 3.0.

SECONDARY OUTCOMES:
Disease free survival | At end of trial- up to 3 years in follow up
Clinical response rate | 4-6 weeks after completion of chemoradiotherapy
R0 resection rate | One week after the operation
Number of Participants who withdraw the treatment | Within the first 84 days after the start of chemoradiotherapy
Perioperative complication | Within the first 90 days after the start of surgery
Pathological complete response rate | One week after the operation
Health Related Quality of Life | Within the first 84 days after the start of chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, Ph.D., M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Wei C, Tucker SL, Myles B, Palmer M, Hofstetter WL, Swisher SG, Ajani JA, Cox JD, Komaki R, Liao Z, Lin SH. Predictors of postoperative complications after trimodality therapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):885-91. doi: 10.1016/j.ijrobp.2013.04.006. PMID 23845841
- [Result] Bhansali MS, Vaidya JS, Bhatt RG, Patil PK, Badwe RA, Desai PB. Chemotherapy for carcinoma of the esophagus: a comparison of evidence from meta-analyses of randomized trials and of historical control studies. Ann Oncol. 1996 Apr;7(4):355-9. doi: 10.1093/oxfordjournals.annonc.a010601. PMID 8805926
- [Result] Arnott SJ, Duncan W, Gignoux M, Hansen HS, Launois B, Nygaard K, Parmar MK, Rousell A, Spilopoulos G, Stewart G, Tierney JF, Wang M, Rhugang Z; Oeosphageal Cancer Collaborative Group. Preoperative radiotherapy for esophageal carcinoma. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD001799. doi: 10.1002/14651858.CD001799.pub2. PMID 16235286
- [Result] Sjoquist KM, Burmeister BH, Smithers BM, Zalcberg JR, Simes RJ, Barbour A, Gebski V; Australasian Gastro-Intestinal Trials Group. Survival after neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal carcinoma: an updated meta-analysis. Lancet Oncol. 2011 Jul;12(7):681-92. doi: 10.1016/S1470-2045(11)70142-5. Epub 2011 Jun 16. PMID 21684205
- [Result] Mariette C, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Robb WB, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF. Surgery alone versus chemoradiotherapy followed by surgery for stage I and II esophageal cancer: final analysis of randomized controlled phase III trial FFCD 9901. J Clin Oncol. 2014 Aug 10;32(23):2416-22. doi: 10.1200/JCO.2013.53.6532. Epub 2014 Jun 30. PMID 24982463
- [Result] Kushida T, Nohara S, Yoshino K, Fujiwara D, Ouchi K, Amano T, Isayama F, Tomita N, Iwanuma Y, Sasai K, Tsurumaru M, Kajiyama Y. Utility of weekly docetaxel combined with preoperative radiotherapy for locally advanced esophageal cancer from pathological analysis. Dis Esophagus. 2014 May-Jun;27(4):368-73. doi: 10.1111/dote.12105. Epub 2013 Jul 19. PMID 23865505
- [Result] Zanoni A, Verlato G, Giacopuzzi S, Weindelmayer J, Casella F, Pasini F, Zhao E, de Manzoni G. Neoadjuvant concurrent chemoradiotherapy for locally advanced esophageal cancer in a single high-volume center. Ann Surg Oncol. 2013 Jun;20(6):1993-9. doi: 10.1245/s10434-012-2822-4. Epub 2012 Dec 29. PMID 23274533
- [Result] Pasini F, de Manzoni G, Zanoni A, Grandinetti A, Capirci C, Pavarana M, Tomezzoli A, Rubello D, Cordiano C. Neoadjuvant therapy with weekly docetaxel and cisplatin, 5-fluorouracil continuous infusion, and concurrent radiotherapy in patients with locally advanced esophageal cancer produced a high percentage of long-lasting pathological complete response: a phase 2 study. Cancer. 2013 Mar 1;119(5):939-45. doi: 10.1002/cncr.27822. Epub 2012 Nov 16. PMID 23165781
- [Result] Ruhstaller T, Widmer L, Schuller JC, Roth A, Hess V, Mingrone W, von Moos R, Borner M, Pestalozzi BC, BalmerMajno S, Koberle D, Terraciano L, Schnider A, Bodis S, Popescu R; Swiss Group for Clinical Cancer Research (SAKK). Multicenter phase II trial of preoperative induction chemotherapy followed by chemoradiation with docetaxel and cisplatin for locally advanced esophageal carcinoma (SAKK 75/02). Ann Oncol. 2009 Sep;20(9):1522-1528. doi: 10.1093/annonc/mdp045. Epub 2009 May 22. PMID 19465425
- [Result] Lin SH, Wang L, Myles B, Thall PF, Hofstetter WL, Swisher SG, Ajani JA, Cox JD, Komaki R, Liao Z. Propensity score-based comparison of long-term outcomes with 3-dimensional conformal radiotherapy vs intensity-modulated radiotherapy for esophageal cancer. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1078-85. doi: 10.1016/j.ijrobp.2012.02.015. Epub 2012 Aug 3. PMID 22867894